CLINICAL TRIAL: NCT04959864
Title: Double-Blind Randomized Controlled Trial Evaluating the Efficacy of the Food Supplement Isitol® Versus Placebo on the Rate of Abnormal Sperm DNA Fragmentation
Brief Title: Efficacy Study of a Food Supplement With Myo-inositol, N-Acetyl-Cystein, Zinc and Vitamins on Sperm DNA Fragmentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GYNOV (Industry)
Collaborators: Laboratoire Drouot (Unknown)
Responsible Party: Sponsor-Investigator, GYNOV, Chief Executive Officer, GYNOV
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-A02402-37
Record Dates: First submitted 2021-06-23; First posted 2021-07-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Male Infertility
Keywords: Spermatozoa; DNA Fragmentation; Chromatin Condensation; Food supplement; TUNEL
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: The randomization scheme is 1 : 1 (treated with food supplement vs placebo). The different treatments (2) have been anonymized, a randomization list is used to assign an anonymous box number (5 random numbers) according to the patient's order of inclusion. Only the promoter is aware of the assignment of the randomization number with which treatment it corresponds.
Who Masked: Participant, Care Provider
Masking Description: The randomization scheme is 1 : 1 (treated with food supplement vs placebo). The different treatments (2) have been anonymized, a randomization list is used to assign an anonymous box number (5 random numbers) according to the patient's order of inclusion. Only the promoter is aware of the assignment of the randomization number with which treatment it corresponds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isitol® (Food supplement treated group) (Experimental): 36 eligible males between 20 and 45 yo. (included limits) will take 1 sachet of Isitol® per day during 16 (± 2) weeks. The sachet of powder is to dissolve in a glass of water or directly in mouth.
  1 sachet of Isitol® (2,1g) contains 1000 mg of myo-inositol, 300 mg of N-acetyl-cysteine, 150 % of the Nutritional Reference Values (NRV) in zinc and 100 % of the NRV: in vitamins B2, B3, B6, B9 and E.
  Interventions: Dietary Supplement: Isitol®
- Placebo treated group (Placebo Comparator): 36 eligible males between 20 and 45 yo. (included limits) will take 1 sachet of placebo per day during 16 (± 2) weeks. The sachet of powder is to dissolve in a glass of water or directly in mouth.
  1 sachet of placebo (2,1g) contains only excipients used in Isitol® and excipients to get similar organoleptic aspect (maltodextrin, sucralose, silicon dioxide, magnesium carbonate, citric acid and beta-carotene).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Isitol® — 1 sachet of Isitol® (2,1g) contains :
  * 1000 mg of myo-inositol ;
  * 300 mg of N-acetyl-cystein ;
  * 48.5 mg of zinc citrate (equivalent zinc pure element : 15 mg) ;
  * 35 mg of D-a-tocopherol (equivalent vitamin E pure element : 12 mg) ;
  * 16 mg of vitamin B3 ;
  * 1.8 mg of pyridoxin hydrochloride (equivalent vitamin B6 pure element : 1.4 mg) ;
  * 1.4 mg of vitamin B2 ;
  * 0.37 mg of (6S)-5-methyltetrahydrofolic acid, glucosamine salt (equivalent vitamin B9 pure element : 0.2 mg).
  Sachets are packaged in box of 30.
  Arms: Isitol® (Food supplement treated group)
Other: Placebo — 1 sachet of placebo (2,1g) contains :
  * 1765.1 of maltodextrin ;
  * 300 mg of magnesium carbonate ;
  * 40 mg of citric acid ;
  * 5.3 mg of beta-carotene ;
  * 2.16 mg of silicon dioxide ;
  * 1.44 mg of sucralose.
  Sachets are packaged in box of 30.
  Arms: Placebo treated group

SUMMARY:
In industrialised countries, it is estimated that about 15% of couples who wish to have a child are currently facing infertility problems, of which, in half of the cases, an anomaly in sperm quality or at least a factor of male origin is identified. The evaluation of sperm quality in males is based, for the most part, on the micro and macroscopic examination of various parameters (concentration, motility, physical abnormalities of the spermatozoa, etc.). Nevertheless, an increasing number of scientific studies have shown that the quality of sperm DNA, and in particular its fragmentation rate, is also associated with a lower fertilisation rate. The integrity of sperm DNA may be affected by an imbalance in the Red/Ox balance leading to uncompensated oxidative stress, and could be restored or improved by dietary hygiene measures and the consumption of specific dietary products. The ISITOL clinical study aims to evaluate the efficacy of a dietary supplement specifically formulated to target the various issues associated with male infertility, and in particular to contribute to the improvement of the sperm DNA fragmentation rate. The efficacy of the dietary supplement Isitol® (GYNOV SAS) on sperm DNA fragmentation rate and other secondary parameters is being evaluated through a single-centre, prospective, randomised, double-blind, interventional vs. placebo clinical study being conducted in France at Laboratoire Drouot (21 Rue Drouot - 75009 Paris - France) and led by Dr. Nino-Guy Cassuto. A total of 72 men aged between 20 and 45 years, with sperm DNA fragmentation rate ≥ 30% and with negative semen culture are recruited. The recruited patients were randomized in a 1:1 scheme into 2 groups (Isitol® treated vs placebo treated).

[Results to be reported later]

DETAILED DESCRIPTION:
Infertility is generally defined as a partner's failure to conceive after at least 12 months off contraception and is steadily increasing worldwide. In industrialised countries, it is estimated that around 15% of couples who wish to have a child are now facing it, and in half of the cases, an abnormality in sperm quality or at least a male factor is identified.

In males, the measurement of male fertility is mainly based on analyses that assess sperm quality macroscopically (spermiogram, spermocytogram) by evaluating the number, morphology, motility, presence of abnormalities, etc. These indicators are still considered to be the preferred indicators for assessing male fertility.

Nevertheless, since the mid-2000s, numerous in vitro and in vivo studies in humans and animals have shown that the integrity of sperm DNA, assessed by measuring the rate of DNA fragmentation and chromatin decondensation in spermatozoa, could be a relevant parameter in the etiology of male infertility. Furthermore, it has been observed that the rate of sperm DNA fragmentation is inversely correlated with pregnancy rate, success rate of assisted reproductive techniques and embryo quality.

The major identified cause of direct damage to DNA molecules and their possible fragmentation, but also to proteins and cell membranes in spermatozoa is oxidative stress. Unreduced Reactive oxygen species produced in the mitochondria-rich midpiece in excess are susceptible to damage the DNA in the sperm head. Several exogenous factors such as exposure to toxins, smoking, alcohol or unbalanced diet are also associated with promoting oxidative stress.

A fragmentation rate higher than 30% is considered high, it is indicative of altered chromatin and especially associated with a low probability of conceiving naturally or through in vitro techniques.

To resolve this problem and improve the process of spermatogenesis and fertilisation, it is relevant to evaluate the effectiveness of a food supplement (Isitol®), manufactured and marketed by the company Gynov SAS (2B Rue Sauteyron - 33000 Bordeaux - France), which provides myo-inositol and a complex with antioxidant properties based on N-acetyl-cysteine, group B vitamins (B2, B3, B6, B9), vitamin E and zinc.

In addition to providing the nutrients that contribute to a better management of the reactive oxygen species, the food supplement provides myo-inositol, which is essential for the functioning of a wide range of cellular functions. This molecule, related to glucose, is produced in the testis, mainly by Sertoli cells, and is excreted into the seminiferous tubules as a gradient. This gradient contributes to sperm maturation by reducing sperm viscosity and increasing sperm motility. Numerous studies evaluating the impact of myo-inositol have shown a significant improvement in sperm parameters (concentration, motility, morphology) and in particular in the rate of sperm DNA fragmentation.

In order to evaluate the efficacy of this dietary supplement, a single-centre, prospective, randomised, double-blind, interventional vs. placebo clinical study was set up in France at Laboratoire Drouot (21 Rue Drouot - 75009 Paris - France) and directed by Dr. Nino-Guy Cassuto. A total of 72 men aged between 20 and 45 years, with sperm DNA fragmentation rate ≥ 30% and with negative semen culture are recruited. The recruited patients were randomised in a 1:1 design into 2 groups (Isitol® treated vs placebo treated).

The primary hypothesis is that after 16 (± 2) weeks of treatment with the dietary supplement, the expected decrease in sperm DNA fragmentation rate will be ≥ 23% compared to the placebo treated group to validate the efficacy hypothesis. The measurement of the sperm DNA fragmentation rate is performed by TUNEL (Terminal deoxynucleotidyl transferase dUTP (deoxyuridine triphosphate) nick end labeling) method. The secondary objectives are the evaluation of classical sperm parameters (spermiogram, spermocytogram), sperm morphology score, chromatin decondensation rate, sperm red/ox potential, differential expression of 11 specific genes involved in spermatogenesis and/or at different stages of the fertilisation process (AURKA, CCDC60, CCDC88B, etc.)).

[Results to be reported later]

ELIGIBILITY:
Selection Criteria:

* Male patient volunteers aged 20 to 45 years (limits included);
* Socially insured patient receiving benefits from the French Social Security's health branch

Non-Selection Criteria:

* Patients suffering from infertility of infectious or genetic origin, or from a pathology requiring concomitant medical treatment;
* Consumption of dietary supplements during the previous 3 months and during the course of the study;
* Smoking ≥ 5 cigarettes/day;
* Alcoholism ≥ 10 drinks (alcohol standard)/week ;
* Body Mass Index (BMI) not between [19 and 29] (inclusive).
* Occupation at risk of exposure to carcinogenic, mutagenic and toxic agents for reproduction defined according to articles R.4412-2 2°, R.4412-3 and R.4412-60 of the French Labour Code;
* Patient unable to give consent;
* Minors and protected adults, vulnerable persons;
* Patient participating in another clinical research study

Inclusion Criteria:

* Sperm DNA fragmentation rate ≥ 30 %

Exclusion Criteria:

* Positive semen culture

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline sperm DNA fragmentation rate at 4 months | Sperm DNA fragmentation rate is measured at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  Sperm DNA fragmentation rate is assessed by the TUNEL (Terminal deoxynucleotidyl transferase dUTP nick end labeling) method. This method is based on the attachment of fluorochrome-coupled biotin-deoxyuridine (dUDP) complexes to the 3'OH ends of possible DNA fragments. The binding of the complexes to the DNA is catalysed by the enzyme Terminal-deoxynucleotidyltransferase. Spermatozoa with fragmented DNA are detected and their percentage measured directly by in-situ confocal fluorescence microscopy.

SECONDARY OUTCOMES:
Change from baseline nuclear chromatin decondensation of spermatozoa at 4 months | Nuclear chromatin decondensation is measured at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  Nuclear chromatin decondensation is assessed by the aniline blue method and expressed in percentage (%).
Change from baseline semen volume at 4 months | Semen volume is mesured at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  Semen volume is expressed in mL.
Change from baseline semen pH at 4 months | Semen pH is measured at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  Semen pH is expressed without unit, the values ranging from 1 to 14.
Change from baseline semen liquefaction time at 4 months | Semen liquefaction time is mesured at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  When the sample is collected it presents a state of coagulation, and must be liquefied to proceed to its study. Semen liquefaction time is expressed in minutes.
Change from baseline spermiogram total spermatozoa, round cells and polynuclear cells count at 4 months | Cells counts are realised at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  The total number of each cell type is counted and expressed in millions (10^6)/ejaculate. The relative concentrations in spermatozoa, round cells and polynuclear cells are obtained after weighting by sample volume and expressed in millions (10^6)/mL.
Change from baseline spermiogram viability and mobility count at 4 months | Viability and mobility are are evaluated at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  Viability and mobility of spermatozoa is evaluated and expressed in percentage (%).
Change from baseline spermocytogram abnormalities count at 4 months | Spermocytogram abnormalities count is realised at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  Spermocytogram is a microscopic analysis of the ejaculate in order to evaluate the number of sperm morphological abnormalities on each part of the spermatozoon (head, middle piece, flagellum).
Change from baseline spermocytogram isolated flagella and of spermatozoa in cell lysis phase numbers at 4 months | Spermocytogram isolated flagella and of spermatozoa in cell lysis phase count is realised at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  Isolated flagella and spermatozoa in cell lysis phase are counted and expressed in percentage (%).
Change from baseline sperm morphology scoring at 4 months | Sperm morphology scoring is realised at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  The score of sperm morphology is assessed according to Cassuto-Barak classification. Spermatozoa are classified into 3 categories (I,II,III) according to the number and/or localisation of morphological abnormalities. The results are expressed in percentage (%) of each class I, II and III.
Change from baseline semen Red/ox potential at 4 months | Red/ox potential measurement is realised at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  The measurement of the semen Red/Ox potential is performed using the MiOXSYS measuring device (Aytu Bioscience 373 Inverness Parkway - Englewood, CO 80112 USA). This device measures the static oxidation reduction potential (sORP) of a biological sample, in this case human semen. The sORP has been described as an integrated measure of the balance between total oxidative activity (including reactive oxygen species) and total reducing activity. Therefore, the level of oxidative stress (increase in oxidative species and/or decrease in antioxidant activity) can be quantified electrically using an sORP sensor. The result is indicated in mV and the increase in sORP is correlated with an increase in the level of oxidative stress. The relative sORP is obtained after weighting by concentration in spermatozoa and expressed in mV/millions (10^6)/mL.
Change from baseline genes expression (AURKA, CCDC60, CCDC88B, CFAP46, HDAC4, CACNA1C, CACNA1H, CARHSP1, DNAH2, HMGB4, SPATA18) at 4 months | Genes expression measurement is realised at first Visit (V0) and at the last Visit (V2) after 16 +/- 2 weeks of treatment with Isitol or placebo
  The expression level of the AURKA, CCDC60, CCDC88B, CFAP46, HDAC4, CACNA1C, CACNA1H, CARHSP1, DNAH2, HMGB4 and SPATA18 genes in spermatozoa will be measured using an RT-qPCR (Reverse transcriptase quantitative polymerase chain reaction) technique with specific primer pairs. The different mRNAs will be extracted from spermatozoa using an extraction kit (miRNeasy Kit (QIAGEN)). Using primers specific to each of the genes studied, the mRNAs of these genes of interest will be back-transcribed into complementary DNA and then amplified according to a determined number of replication cycles (45 cycles). By measuring the fluorescence intensity in each of the cells, the concentration of complementary DNA is calculated. The relative expression of these different genes is obtained after normalisation using two ubiquitous and constant expression genes.

CONTACTS AND LOCATIONS:
Overall Officials: Nino-Guy Cassuto, PharmD, Principal Investigator — Laboratoire Drouot
Locations (1):
- Laboratoire Drouot, Paris, France

IPD SHARING:
Plan to Share IPD: No